CLINICAL TRIAL: NCT03053609
Title: Association Between Cardiorespiratory and Gastroesophageal Reflux Events in Infants.
Brief Title: Gastroesophageal Reflux and Cardiorespiratory Problems
Acronym: CR-GER
Status: Completed | Type: Observational
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Francesco Cresi, Principal Investigator, University of Turin, Italy
Other Study IDs: apnea-01
Record Dates: First submitted 2017-02-09; First posted 2017-02-15 (Actual); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Gastroesophageal Reflux Disease; Apnea Infants; Desaturation of Blood; Bradycardia
Keywords: gastroesophageal reflux; apnea; bradycardia; desaturation; impedance
MeSH Terms: conditions — Gastroesophageal Reflux; Bradycardia; Apnea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cardiorespiratory and gastroesophageal reflux events often coexist in infants in Neonatal Intensive Care Unit (NICU) thus leading to drugs over-prescription and delayed discharge.

Through cardiorespiratory and pH-impedance monitoring this study aims to evaluate the temporal association between gastroesophageal reflux (GER) and cardiorespiratory (CR) events in a large number of infants with gastroesophageal reflux disease (GERD) and CR symptoms and, whether this association is significant, to clarify the impact of GER on CR events.

DETAILED DESCRIPTION:
This is an observational retrospective study to describe the association between cardiorespiratory (CR) and gastroesophageal reflux (GER) events in infants who underwent synchronized 24h Multichannel Intraluminal Impedance/pH-metry (MII/pH) and CR monitoring for GER disease symptoms and CR events. Data are collected from medical records and database of the University Neonatal Intensive Care Unit of the Sant'Anna-Regina Margherita Children Hospital (Turin).

The symptom association probability (SAP) index is used to identify those infants with significant associations between GER and CR events. In the group of infants with a positive SAP index the differences in reflux characteristics are compared according to whether a reflux preceded or followed a cardiorespiratory event (30 s time window).

ELIGIBILITY:
Inclusion Criteria:

* synchronized MII-pH and cardio-respiratory monitoring lasting more than 12 hours, excluding meal periods;
* exclusive enteral feeding
* parents' informed consent

Exclusion Criteria:

* infectious, genetic, metabolic and neurological diseases
* ventilatory support and/or oxygen supplementation at the time of MII-pH/CR monitoring
* pharmacological therapies with effects on GER or apnoea during the week before MII-pH/CR monitoring

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants admitted to the University Neonatal Intensive Care Unit of the Sant'Anna-Regina Margherita Children Hospital from January 2006 to December 2016 who underwent 24h synchronized pH-impedance and cardiorespiratory monitoring for GER disease symptoms and cardiorespiratory events.
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2006-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
SAP index | calculated throughout 24 hours
  Symptom Association Probability (SAP) between gastroesophageal reflux and cardio-respiratory events. SAP is considered positive if > 95%.

SECONDARY OUTCOMES:
Gastroesophageal reflux frequency | calculated throughout 24 hours
  Reflux event is defined as: a drop of impedance to 50% of the basal value for at least 5 s, starting in the most distal channel and proceeding to one or more proximal channels and followed by a recovery of the impedance baseline values

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Cresi, MD, PhD, Principal Investigator — University of Turin, Italy
Locations (1):
- Ospedale S.Anna di Torino, Torino, (to), Italy

IPD SHARING:
Plan to Share IPD: No